CLINICAL TRIAL: NCT05617612
Title: Neonatal Alloantibodies in Cord Blood for Early Detection of Hemolytic Disease of Newborn
Brief Title: Neonatal Cord Blood Screening for HDN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaaa Abd El-Aleem, Neonatal Alloantibodies in cord blood for early detection of Hemolytic disease of newborn, Assiut University
Other Study IDs: HDN screening
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: HDN - Hemolytic Disease of the Newborn
MeSH Terms: conditions — Erythroblastosis, Fetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the diagnostic efficiency of antibodies screening in cord blood for detection of HDN.

To help finding the antigen negative blood in a timely manner and reduce the morbidities and mortalities of HDN

DETAILED DESCRIPTION:
Hemolytic disease of the newborn (HDN) refers to fetal or neonatal alloimmune hemolysis caused by red blood cell antibodies due to incompatible maternal and fetal or neonatal blood types. A French midwife first described the disorder in 1609; however, it was not until the 1950s when the underlying cause was clarified. The pathogenesis of HDN begins with the attack of fetal red blood cells (RBCs) by maternal antibodies due to incompatibility of maternal and fetal blood. Immunologically, antibody secretion initially starts with Immunoglobulin M (IgM), which cannot cross the placental barrier, but is then followed by isotype switching, which produces Immunoglobulin G (IgG) antibodies. IgG antibodies can cross the placental barrier, and they do so during the second and or subsequent pregnancies, attacking the fetal RBCs and causing hemolysis and associated complications such as Hydrops fetalis and jaundice. HDN can occur due to Rh antigens, most commonly the D antigen, and A,B and O RBCs antigens (ABO) antigens. Rh(D)-HDN has decreased since the introduction of antenatal and postpartum Rh immunoglobulin. Therefore, the prevalence of HDN, nowadays, varies according to blood type incompatibility. ABO incompatibility is the most common cause of HDN and Rh (D) antigen is the second most common cause.[8] Rh (C, c, E, e) antigen incompatibility occurs occasionally. Several other alloantibodies have also been reported to be associated with hemolytic diseases, including Kidd, Diego, Duffy, Kell and Anti-Mur. Minor blood group incompatibility due to blood groups other than Rh(D), although an uncommon cause of neonatal hyperbilirubinemia, has the potential to cause severe hyperbilirubinemia and its sequelae in infants, if left undiagnosed and untreated. Therefore, identification of at-risk cases will help clinicians to reduce neonatal morbidity and will result in better patient management

ELIGIBILITY:
Inclusion Criteria:

* Full term neonates >/= 37 weeks.
* ABO blood compatible mother and neonate

Exclusion Criteria:

* Preterm neonates < 37 weeks.
* ABO incompatibility between mother and neonate

Ages: 1 Day to 3 Days | Sex: All
Age Groups: Child
Study Population: Full term neonates who have ABO blood group compatibility with their mothers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the diagnostic efficiency of antibodies screening in cord blood for detection of HDN | Baseline
  Early detection of HDN through antibodies screening would help finding the antigen negative blood in a timely manner and reduce the morbidities and mortalities

REFERENCES:
- [Background] Lin M, Liu M, Zhang S, Chen C, Wang J. Different Types of Minor Blood Group Incompatibility Causing Haemolytic Disease of Neonates in one of the National Children's Medical Centre in China. J Blood Med. 2021 Jun 25;12:497-504. doi: 10.2147/JBM.S303633. eCollection 2021. PMID 34211305
- [Background] Jackson ME, Baker JM. Hemolytic Disease of the Fetus and Newborn: Historical and Current State. Clin Lab Med. 2021 Mar;41(1):133-151. doi: 10.1016/j.cll.2020.10.009. Epub 2020 Dec 24. PMID 33494881
- [Background] Gupta GK, Balbuena-Merle R, Hendrickson JE, Tormey CA. Immunohematologic aspects of alloimmunization and alloantibody detection: A focus on pregnancy and hemolytic disease of the fetus and newborn. Transfus Apher Sci. 2020 Oct;59(5):102946. doi: 10.1016/j.transci.2020.102946. Epub 2020 Sep 16. PMID 32962917
- [Background] Alaqeel AA. Hyporegenerative anemia and other complications of rhesus hemolytic disease: to treat or not to treat is the question. Pan Afr Med J. 2019 Mar 14;32:120. doi: 10.11604/pamj.2019.32.120.17757. eCollection 2019. PMID 31223410
- [Background] Tewari VV, Kumar A, Singhal A, Pillai N, Prakash A, Varghese J, Kannan V. Evaluation of Rh-Hemolytic Disease in Neonates and Management with Early Intensive Phototherapy in the Neonatal Intensive Care Unit. J Trop Pediatr. 2020 Feb 1;66(1):75-84. doi: 10.1093/tropej/fmz033. PMID 31199484